CLINICAL TRIAL: NCT01759251
Title: Post-marketing Observational Program of Betaserc® (Betahistine Dihydrochloride) to Evaluate Effectiveness in Patients With Vestibular Vertigo in Routine Practice
Brief Title: Effectiveness of Betaserc® (Betahistine Dihydrochloride) in Patients With Vestibular Vertigo in Routine Practice
Acronym: VIRTUOSO
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P13-972
Record Dates: First submitted 2012-12-28; First posted 2013-01-03 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Vertigo
Keywords: Meniere Disease; Betahistine Dihydrochloride; Vertigo
MeSH Terms: conditions — Vertigo; Meniere Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- vestibular vertigo: Patients with vestibular vertigo of known or unknown origin, and for whom the physician has decided to prescribe betahistine dihydrochloride at dose 48 mg/day in accordance with locally approved label

SUMMARY:
The purposes of this international post-marketing observational program is to investigate effectiveness of betahistine dihydrochloride (Betaserc®) tablets and assess the course of vestibular vertigo after treatment discontinuation in population of Russia and Ukraine outpatients suffering from vestibular vertigo in pragmatic clinical settings. Exploratory analyses of results from both participating countries may be expected to provide insights about the subjective circumstances of vestibular vertigo patients in a wider than usual range of gender, underlying ICD-10 diagnosis, national and cultural situations.

DETAILED DESCRIPTION:
A prospective, multicentre, non-interventional, non-randomized, non-controlled, single arm, post-marketing observational program in patients whom betahistine dihydrochloride (Betaserc®) tablets were prescribed in the usual manner at the maximal recommended daily dose of 48 mg in accordance with the locally approved label. Over a program period physician is free to adjust betahistine dihydrochloride dose according to country approved label. Adult outpatients with vestibular vertigo who can be treated with betahistine dihydrochloride as per the locally approved label will be enrolled in the program. The program consists of an observational treatment period (up to 2 months) and a follow-up period (up to 2 months, for evaluation of the course of vestibular vertigo after treatment completion).

ELIGIBILITY:
Inclusion Criteria

* Male or female 18 years and older.
* Patients with vestibular vertigo of known or unknown origin, and for whom the physician has decided to prescribe 48 mg of betahistine dihydrochloride (Betaserc®) in accordance with locally approved label.
* Patients who are willing and able to provide authorization to the investigator to use and/or disclose personal and/or health data.
* Patients who started betahistine dihydrochloride (Betaserc®) therapy not more than 5 days priory to sign Patient Authorization (Consent) for Use/Disclosure of Data.

Exclusion Criteria

* Patients with any condition which, in the opinion of the Investigator, makes the patient unsuitable for inclusion based on clinical judgment.
* Labeled contraindications of betahistine dihydrochloride (Betaserc®) treatment.
* Patients with middle or inner ear infection.
* Patient with psychiatric disorders, significant neurological disorder or spinal cord damage.
* Patients receiving any other agents for peripheral vestibular vertigo such as diuretics, transtympanic gentamycin, cinnarizine, competitive antagonist of histamine, blocking H1- histamine receptors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients with vestibular vertigo
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal Berrou, MD, Study Director — Abbott
Locations (24):
- Russia (15):
  - Site reference ID 89414, Belgorod
  - Research facility ID ORG-000838, Irkutsk
  - Site reference ID 89433, Kazan'
  - Site reference ID 89454, Moscow
  - Site reference ID 89419, Moscow
  - Research facility ID ORG-000837, Moscow
  - Site reference ID 94374, Moscow
  - Site reference ID 89416, Moscow
  - Site reference ID 89435, Novosibirsk
  - Research facility ID ORG-000841, Odintsovo
  - Site reference ID 89453, Rostov-on-Don
  - Site reference ID 89456, Saint Petersburg
  - Site reference ID 89418, Saratov
  - Site reference ID 89415, Ufa
  - Site reference ID 89455, Volgograd
- Ukraine (9):
  - Research facility ID ORG-000345, Donetsk
  - Site reference ID 93715, Ivano-Frankivsk
  - Site reference ID 93713, Kharkiv
  - Site reference ID 93454, Kiev
  - Site reference ID 93475, Mykolaiv
  - Site reference ID 93714, Sevastopol
  - Site reference ID 93474, Simferopol
  - Site reference ID 95738, Zaporizhzhia
  - Site reference ID 93455, Zaporizhzhia

RESULTS

PARTICIPANT FLOW:
Period: 30 Days Treatment Period
Arm/Group | Vestibular Vertigo
Started | 309
Completed | 305
Not Completed | 4
Period: 60 Days Treatment Period
Arm/Group | Vestibular Vertigo
Started | 305
Completed | 305
Not Completed | 0
Period: Follow-up Period
Arm/Group | Vestibular Vertigo
Started | 305
Completed | 305
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with vestibular vertigo of known or unknown origin, and for whom the physician has decided to prescribe 48 mg of Betaserc® in accordance with locally approved label.
Arm/Group | Vestibular Vertigo
Number analyzed (Participants) | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220
  Male | 89
Region of Enrollment [Number; unit: participants]
  Ukraine | 102
  Russian Federation | 207

OUTCOME MEASURES:

1. Primary Outcome: Scale for Vestibular Vertigo Severity Level and Clinical Response Evaluation (SVVSLCRE)
Description: Number of patients with clinical response on treatment determined with SVVSLCRE
Time Frame: Up to 2 months
Population: 60 days treatment group
Measure: Number; unit: participants
Arm/Group | Vestibular Vertigo
Number analyzed (Participants) | 305
participants
  excellent | 43
  very good | 79
  good | 104
  moderate | 61
  no change | 15
  worsening | 3

2. Secondary Outcome: Change of the Patient's Clinical Conditions of Vestibular Vertigo From Baseline to the End of Observational Treatment Period
Description: determined with the Scale for Vestibular Vertigo Severity Level and Clinical Response Evaluation (SVVSLCRE)
Time Frame: From Day 0 to 2 months
Reporting Status: Not Posted

3. Secondary Outcome: Change of Vestibular Vertigo Attacks Frequency From Baseline to the End of Observational Treatment Period
Time Frame: From Day 0 to 2 months
Reporting Status: Not Posted

4. Secondary Outcome: Change of Vestibular Vertigo Attacks Frequency From the End of Observational Treatment Period to the End of Follow-up Period
Time Frame: From 2 months to 4 months
Reporting Status: Not Posted

5. Secondary Outcome: Overall Clinical Response Assessed by Physician
Description: determined with a four-point-scale, where 4 = excellent, 3 = good, 2 = fair, and 1 = poor.
Time Frame: up to 2 months
Reporting Status: Not Posted

6. Secondary Outcome: Overall Clinical Response Assessed by Patient
Description: determined with a four-point-scale, where 4 = excellent, 3 = good, 2 = fair, and 1 = poor.
Time Frame: up to 2 months
Reporting Status: Not Posted

7. Secondary Outcome: Clinical Response as Improvement of Vertigo Associated Symptoms Evaluated by Physician
Description: vertigo associated symptoms: tinnitus, hearing loss, nausea, vomiting, faintness and headache; determined with a four-point-scale, where 4 = excellent, 3 = good, 2 = fair, and 1 = poor.
Time Frame: up to 2 months
Reporting Status: Not Posted

8. Secondary Outcome: Clinical Response as Improvement of Vertigo Associated Symptoms Evaluated by Patient
Description: as for outcome 7
Time Frame: up to 2 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Serious adverse events will be reported to Abbott from the time the physician obtains the patient's authorization to use and disclose information (or the patient's informed consent) until 30 days following the intake of the last dose of physician-prescribed treatment.
Arm/Group | Vestibular Vertigo
Serious Adverse Events (participants affected / at risk) | 0/309
Other Adverse Events (participants affected / at risk) | 0/309

LIMITATIONS AND CAVEATS:
4 patients had a treatment exposure of 30 days. No subgroup analyses were performed as the majority of patients had 60 days treatment with Betaserc®.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall not publish /present the results without Abbott's prior written consent. In the event that applicable law permits Investigator to publish or present results without Abbott's prior written consent, Investigator shall provide Abbott with a complete copy of such publication or presentation at least 60 days prior to submission for publication or presentation and Investigator shall reasonably consider all comments which Abbott may provide regarding such publication or presentation.